CLINICAL TRIAL: NCT01163409
Title: Acupuncture and Physical Activity in Patients With Fibromyalgia
Brief Title: Exercise, Acupuncture and Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo (Other)
Responsible Party: Clóvis Artur Almeida da Silva/ MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: exercisefibro
Record Dates: First submitted 2010-06-09; First posted 2010-07-15 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2010-06

CONDITIONS: Fibromyalgia; Juvenile
Keywords: juvenile fibromyalgia; acupuncture; exercise training
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise; Sex Education; Psychotherapy; Acupuncture Therapy; Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- acupuncture (Experimental): will be made with classic acupuncture needling in traditional points, surpassing the skin
  Interventions: Procedure: acupuncture; Procedure: Exercise, Acupuncture and Fibromyalgia
- sham acupuncture (Experimental): sham acupuncture will be done through a needle and a plastic device attached to skin in traditional acupuncture points.
  Interventions: Procedure: Exercise, Acupuncture and Fibromyalgia
- exercise training resistance and aerobic (Experimental): Aerobic exercise for 1 hour and resistance exercises for major muscle groups.
  Interventions: Procedure: exercise training; Procedure: Exercise, Acupuncture and Fibromyalgia
- healthy lifestyle (No Intervention): Group 4 - will be the control group who receive follow-up and recommendation for physical activity, but without any intervention supervised.
  Interventions: Procedure: Exercise, Acupuncture and Fibromyalgia

INTERVENTIONS:
Procedure: exercise training — exercise training comprises aerobic and strength training
  Other Names: Multidisciplinary treatment including medication; Family education; Psychotherapy; Interventions to reduce pain; Improve sleep quality.
  Arms: exercise training resistance and aerobic
Procedure: acupuncture — acupuncture involves two sessions per week, during 14 weeks.
  Other Names: Systematic study of physical activity and acupuncture have stimulated
  Arms: acupuncture
Procedure: Exercise, Acupuncture and Fibromyalgia — Set of real acupuncture treatment and supervised aerobic exercise have better efficacy in pediatric patients with fibromyalgia versus treatment with sham acupuncture and supervised aerobic exercise, as well as treatment versus combination with aerobic exercise and resistance exercise the major muscle groups, both supervised versus group control, we just get guidance for physical activity.
  Other Names: Assess pain reduction; Improvement in quality of life in children and adolescents; Compare four treatment groups

SUMMARY:
Set of real acupuncture treatment and supervised aerobic exercise have better efficacy in pediatric patients with fibromyalgia versus treatment with sham acupuncture and supervised aerobic exercise, as well as treatment versus combination with aerobic exercise and resistance exercise the major muscle groups, both supervised versus group control, who just get guidance for physical activity.

DETAILED DESCRIPTION:
Fibromyalgia syndrome is a chronic musculoskeletal pain of unknown etiology. It is characterized by diffuse musculoskeletal pain or painful specific sites, usually accompanied by sleep disorders, fatigue, morning stiffness, chronic headaches, mental disorders and functional bowel. The diagnosis is essentially clinical, with no abnormal laboratory and radiological features Physical exercises are part of the treatment of fibromyalgia, but does not report studies in children. In general children with fibromyalgia are encouraged to a multidisciplinary treatment including medication, family education and child graduated aerobic exercise, psychotherapy, interventions to reduce pain, stress and improve sleep quality. To date no studies in medical literature with the use of acupuncture and supervised physical activity in juvenile fibromyalgia.

The significant sample of this disease, our recent publications in this research and the lack of systematic study of physical activity and acupuncture have stimulated this research. Assess pain reduction and improvement in quality of life in children and adolescents with juvenile fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile fibromyalgia diagnosis
* Age between ten to seventeen years and eleven months

Exclusion Criteria:

* Previous treatment with acupuncture;
* Treatment with psychotherapy, exercise training, use of antidepressant and anti-inflammatory drugs in the last month;
* Inflammatory diseases, hypothyroidism and hyperthyroidism

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
pain | 14 weeks
  Clinical evaluation of pain is made by a general questionnaire for pain and overall evaluation of the patient / family and professional by the Visual Analogue Scale. There will be pain as described in 18 points for fibromyalgia, using as instrument the pressure algiômetro Fischer, settling myalgic index.

SECONDARY OUTCOMES:
quality of life | 14 weeks
  Functional assessment of quality of life will be made by the Childhood Health Assessment Questionnaire (CHAQ) of pediatric Peds QL questionnaire that will be answered by the patients and their parents in age groups: 9-12 years and 13-18 years.
strength | 14 weeks
  will be assessed by means of 1-RM test

CONTACTS AND LOCATIONS:
Overall Officials: Clóvis AA Silva, M.D, Ph.D, Principal Investigator — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Magda Maria Maia, São Paulo, São Paulo
  - University of Sao Paulo, São Paulo, São Paulo